CLINICAL TRIAL: NCT02369666
Title: Effects of 4-weeks Ingestion of LycoRed 40051 Product on Exercise-Induced Inflammation, Muscle Damage, and Oxidative Stress in Endurance Runners
Brief Title: LycoRed 40051 Product as a Countermeasure to Exercise Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: LycoRed Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-0093
Record Dates: First submitted 2015-01-30; First posted 2015-02-24 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Inflammation
Keywords: Inflammation; Lycopene; Exercise
MeSH Terms: conditions — Inflammation; Motor Activity | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LycoRed (code 40051) product (Experimental): Dietary supplement, LycoRed (code 40051) product, experimental: Mixture of tomato-based carotenoids and phytochemicals in medium chain triglycerides (MCT). One capsule each day with the morning meal, for 4 weeks.
  Interventions: Dietary Supplement: LycoRed (code 40051) product; Dietary Supplement: Placebo
- Placebo (Placebo Comparator): Dietary supplement placebo: Only MCT oil. One capsule each day with the morning meal, for 4 weeks.
  Interventions: Dietary Supplement: LycoRed (code 40051) product; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: LycoRed (code 40051) product — Mixture of tomato lycopene and carotenoids.
Dietary Supplement: Placebo — Contains MCT oil.

SUMMARY:
The primary purpose of this study is to determine if 4-weeks ingestion of LycoRed (code 40051) product containing a mixture of tomato extract with carotenoids and phytochemicals by endurance runners attenuates inflammation, muscle damage and soreness, and oxidative stress during 24 hours recovery from a 2-h running bout.

DETAILED DESCRIPTION:
STUDY DESIGN

* Randomized-crossover, double-blind, placebo-controlled study, with N=20 endurance runners. (May start with up to 26 subjects to ensure that 20 subjects complete all study requirements). Subjects will ingest the supplement for 4 weeks prior to running 2 hours at high intensity, washout for 2 weeks, crossover and ingest the supplement for 4 weeks prior to running 2 hours at high intensity.
* 2 arms: LycoRed (code 40051) product and placebo.
* During the 3-day period prior to each running session, subjects will taper exercise training and ingest a moderate-carbohydrate diet using a food list restricting high fat foods and visible fats. Subjects will record all food and beverage intake during the 3-day period, with macro- and micro-nutrient intake assessed using the Food Processor dietary analysis software system (ESHA Research, Salem, OR).
* Exercise protocol: Subjects (overnight fasted) will run on laboratory treadmills at 70% VO2max (~marathon race pace) for 1.5 hours followed by 30 minutes of downhill running (10%) at the same intensity. The downhill running portion will induce delayed onset of muscle soreness (DOMS). The run sessions will occur at 7:00-9:00 am.
* Blood samples will be collected pre- and post-4 weeks supplementation, and immediately post-, 1-h post-, and 24-h post-exercise. DOMS will be measured using a 10-point Likert scale at each blood sampling time point.

STUDY PERFORMANCE

* Male and female endurance runners in the Kannapolis/Charlotte, NC metropolitan area will be recruited through mass advertising and direct email messages. Runners will also be recruited during the Expo event the day before the Charlotte Marathon.
* Study duration is 10 weeks, with 6 visits to the ASU-NCRC Human Performance Lab, two exercise sessions, and 10 blood samples.
* Visit 1: 0-week, pre-study, baseline testing and orientation, early morning; provide blood sample (overnight fasted). Subjects will sign the consent form, fill in the ACSM/AHA screening questionnaire, and complete a training history questionnaire. Subjects will be tested for VO2max (treadmill graded exercise test with metabolic measurement), and body composition (BodPod). Subjects will be given instructions for taking the supplements, and initiate supplementation (4-weeks) (with capsules contained in supplement trays to improve compliance). Subjects will be asked to maintain their normal training schedules, and will record weekly training distances in a log.
* Visit 2: 4-weeks, ~7:00 am, overnight fasted; provide blood pre- and post-running for 2 h (70% VO2max), and 1-h post run.
* Visit 3: ~7:00 am, overnight fasted, 24-h post-run: provide blood sample. Start 2-week washout period.
* Visit 4: 6-weeks, provide blood sample (~7:00 am, overnight fasted), crossover to opposite study arm, and start 4-week supplementation.
* Visit 5: 10-weeks, (~7:00 am, overnight fasted), provide blood pre- and post-running for 2 h (70% VO2max), and 1-h post run.
* Visit 6: 24-h post-run (~7:00 am, overnight fasted), provide final blood sample.

INVESTIGATIONAL PRODUCTS

* LycoRed (code 40051) product with mixture of selected carotenoids and phytochemicals in medium chain triglycerides (MCT).
* Placebo: Each softgel will be identical looking, containing the vehicle of MCT oil with all active ingredients removed.
* One serving (1 capsule) of the supplement will be consumed daily during the morning meal.

PRIMARY ENDPOINT

• Oxidative stress biomarkers

SECONDARY ENDPOINTS

* Inflammation biomarkers
* Muscle damage biomarkers
* Plasma lycopene, phytofluene, and phytoene
* Oxidative capacity

ELIGIBILITY:
Inclusion Criteria:

* Male or female endurance runner (ages 18 to 45).
* Compete in long distance road races and are capable of running on a treadmill at marathon race pace for two hours (including 30 min of downhill running). Note: Preference will be given to runners who have completed a half-marathon or greater distance race in the previous year.
* At "low risk" status for cardiovascular disease (as determined with the screening questionnaire).
* Agree to train normally, stay weight stable, and avoid the use of large-dose vitamin/mineral supplements (above 100% of recommended dietary allowances), herbs, and all medications during the project.
* Agree to taper exercise prior to each of the two lab running sessions as if preparing for a long distance race.

Exclusion Criteria:

* Inability to comply with study requirements.
* Any other concurrent condition which, in the opinion of the primary investigator (PI), would preclude participation in this study or interfere with compliance.
* Weigh less than 110 pounds.
* Current, active history of coronary heart disease, stroke, cancer, diabetes, rheumatoid arthritis, high blood pressure, kidney disease, liver disease, blood disease, hormonal disease, or metabolic disease.
* History of cancer in the 5 years prior to the screening visit (except skin or cervical cancer that was successfully treated).
* Current use of any type of medication (or unwillingness to stop use of over-the-counter medications two weeks before the start of the study).
* Use of any 'recreational substance' whether legal or illegal, by prescription or over the counter.
* Pregnant or nursing, or planning to be pregnant or nursing during the study.
* Use of vitamin/antioxidant supplements within 4 weeks prior to starting the study. For subjects using vitamin/antioxidant supplements, a 4-week wash out will be required prior to starting the study.
* Unwilling to follow dietary guidelines from the screening visit through the final visit as follows:
* no more than an average of 2 servings*/week of lycopene-rich foods (e.g. tomatoes and tomato products, including all sauces containing tomatoes that are contained in pizza, soups, etc., ketchup, vegetable juice with tomato, French salad dressing, mango, guava, watermelon, papaya, red grapefruit).
* no more than an average of 5 servings*/day of vegetables and fruit
* avoidance of antioxidant vitamin, mineral or herbal supplements including, but not limited to vitamin C, vitamin E, flavonoids, carotenoids, selenium, etc.
* Consumption of more than an average of 2 units of alcohol daily.**
* Known allergy to tomatoes or citrus fruits.
* Following any special diet including, but not limited to liquid, high or low protein, raw food, vegetarian or vegan, etc. (Subjects should normally consume mixed diets).
* Current use of muscle enhancing supplements such as HMB, ATP and other similar muscle building agents.
* Current use of use of sodium bicarbonate or medications containing sodium bicarbonate such as Alka-Seltzer.
* Recent history of musculoskeletal trauma (fracture, strain, sprain, etc.) that has not fully healed prior to baseline testing.
* Planning to have surgery during the study.

  * For the purpose of this study one serving of vegetables or fruit is defined as: Vegetables
* 1 c raw leafy vegetable; ½ c cut-up raw or cooked vegetable; ½ c vegetable juice Fruit
* 1 med fruit; ¼ c dried fruit; ½ c fresh, frozen, or canned fruit; ½ c fruit juice

  * For the purpose of this study, one unit of alcohol is defined as 12 oz (400 ml) of beer, 6 oz (200 ml) of wine or 1.5 oz (50 ml) of hard spirits.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in exercise-induced oxidative stress | baseline and 4 weeks/pre-exercise, immediately post-exercise, 1-hour post-exercise, 24-hours post-exercise
  F2-isoprostanes.

SECONDARY OUTCOMES:
Change in plasma carotenoids, composite (lycopene, phytofluene, and phytoene) | baseline and 4 weeks/pre-exercise, immediately post-exercise, 1-hour post-exercise, 24-hours post-exercise
  Indicators of tomato paste product ingestion
Change in exercise-induced muscle damage marker | baseline and 4 weeks/pre-exercise, immediately post-exercise, 1-hour post-exercise, 24-hours post-exercise
  Creatine kinase
Change in exercise-induced muscle damage marker | baseline and 4 weeks/pre-exercise, immediately post-exercise, 1-hour post-exercise, 24-hours post-exercise
  Myoglobin
Change in exercise-induced inflammation | baseline and 4 weeks/pre-exercise, immediately post-exercise, 1-hour post-exercise, 24-hours post-exercise
  C-reactive protein
Change in exercise-induced inflammation, composite | baseline and 4 weeks/pre-exercise, immediately post-exercise, 1-hour post-exercise, 24-hours post-exercise
  six inflammatory cytokines, MSD panel (plasma IL-6, IL-8, IL-10, TNF-α, G-CSF, MCP-1)
Change in exercise-induced oxidative stress | baseline and 4 weeks/pre-exercise, immediately post-exercise, 1-hour post-exercise, 24-hours post-exercise
  Protein carbonyls
Change in exercise-induced oxidative stress | baseline and 4 weeks/pre-exercise, immediately post-exercise, 1-hour post-exercise, 24-hours post-exercise
  red blood cell glutathione
Change in oxidative capacity | baseline and 4 weeks/pre-exercise, immediately post-exercise, 1-hour post-exercise, 24-hours post-exercise
  FRAP (Ferric Reducing Ability of Plasma)

CONTACTS AND LOCATIONS:
Overall Officials: David C. Nieman, DrPH, Principal Investigator — Professor
Locations (1):
- Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States

REFERENCES:
- [Result] Ahmed M, Henson DA, Sanderson MC, Nieman DC, Gillitt ND, Lila MA. The protective effects of a polyphenol-enriched protein powder on exercise-induced susceptibility to virus infection. Phytother Res. 2014 Dec;28(12):1829-36. doi: 10.1002/ptr.5208. Epub 2014 Aug 2. PMID 25088029
- [Result] Nieman DC, Shanely RA, Luo B, Meaney MP, Dew DA, Pappan KL. Metabolomics approach to assessing plasma 13- and 9-hydroxy-octadecadienoic acid and linoleic acid metabolite responses to 75-km cycling. Am J Physiol Regul Integr Comp Physiol. 2014 Jul 1;307(1):R68-74. doi: 10.1152/ajpregu.00092.2014. Epub 2014 Apr 23. PMID 24760997
- See also: North Carolina Research Campus — http://transforming-science.com/